CLINICAL TRIAL: NCT02626143
Title: Effect of Feeding Mode on Infant Growth and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Instituto de Nutricion y Tecnologia de los Alimentos (INTA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 6029
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Infant Nutrition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational nutrient-rich whey protein formula (Experimental)
  Interventions: Other: Investigational nutrient-rich whey protein formula
- Cow's milk based formula (Active Comparator)
  Interventions: Other: Cow's milk based formula
- Breast milk (No Intervention)

INTERVENTIONS:
Other: Investigational nutrient-rich whey protein formula
  Arms: Investigational nutrient-rich whey protein formula
Other: Cow's milk based formula
  Arms: Cow's milk based formula

SUMMARY:
This study is intended to compare growth, nutritional status, and brain development in children fed an Investigational cow's milk based formula containing a nutrient-rich whey protein, a standard cow's milk based formula, or fed exclusively breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, 0-120 days of age at study entry
* Term infant with birth weight of 2500 to 4500 grams
* Exclusively feed infant formula or exclusively feeding breast milk
* Signed informed consent

Exclusion Criteria:

* History of underlying metabolic or chronic disease, congenital malformation, or immunocompromised.
* Feeding difficulties or formula intolerance
* Receiving complementary feedings

Ages: 0 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 582 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Body weight | 24 months
Auditory Event-related Potential | 24 months
Body length | 24 months
Head circumference | 24 months

SECONDARY OUTCOMES:
Dietary Intake | 24 months
Medically confirmed adverse events | 24 months
Body Composition: Air Displacement Plethysmography | 6 months
Body Composition: Deuterium Dilution | 12 and 24 months
Blood sample: Micronutrient status | 24 months
Blood sample: Metabolic markers | 24 months
Bayley Scales of Infant and Toddler Development | 12 months
Sleep measures (Amount of time awake & asleep in a 7-day period) | 24 months
Language development: Native3 Phoneme Repertory | 12 months
Language development: Word Discovery | 10 months
Language development: Rule Inference | 10 months
Language development: MacArthur Communicative Development Inventory | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol Lynn Berseth, MD, Study Director — Mead Johnson Nutrition
Locations (1):
- Instituto de Nutricion y Tecnologia de los Alimentos, Santiago, Chile

REFERENCES:
- [Derived] Toro-Campos R, Algarin C, Peirano P, Pena M, Murguia-Peniche T, Wu SS, Uauy R. Effect of feeding mode on infant growth and cognitive function: study protocol of the Chilean infant Nutrition randomized controlled Trial (ChiNuT). BMC Pediatr. 2020 May 18;20(1):225. doi: 10.1186/s12887-020-02087-9. PMID 32423392